CLINICAL TRIAL: NCT04587024
Title: A Pilot Study of mDOT for Immunosuppressant Adherence in Solid Organ Transplant Recipients
Brief Title: A Study of mDOT for Immunosuppressant Adherence in Solid Organ Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB00257447
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Medication Adherence; Liver Transplantation; Kidney Transplantation
MeSH Terms: conditions — Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth intervention (Other): mHealth intervention
  Interventions: Other: mHealth intervention
- standard of care (Placebo Comparator): post-transplant standard of care
  Interventions: Other: standard of care

INTERVENTIONS:
Other: mHealth intervention — Subjects will receive mHealth direct observation of therapy for 12 weeks
  Arms: mHealth intervention
Other: standard of care — Subjects will receive standard of care observation for 12 weeks
  Arms: standard of care

SUMMARY:
In solid organ transplant recipients, poor adherence to immunosuppressant medications carries the risk of graft rejection (needing a new transplant), post-transplant complications, and increased healthcare costs. Additionally, nonadherence to immunosuppressant medications is imperative to short- and long-term outcomes. The rate of nonadherence in this population varies vastly. Because of lacking objective and accurate nonadherence measurements, both to immunosuppressant drugs and medical indications, the true implications and prevalence of nonadherence is not yet well understood. Therefore, investigators believe that mobile health (mHealth) technology has the potential to allow clinicians and researchers to more comprehensively address and understand nonadherence in solid organ transplant recipients. The aim of this study is to conduct a randomized control trial to compare medication adherence among liver and kidney transplant patients who use the mHealth system against controls who do not.

DETAILED DESCRIPTION:
1. STUDY OBJECTIVES 1.1 Primary Objective To compare medication adherence of solid organ transplant recipients, specifically liver and kidney transplants, using the mobile DOT (mDOT) application (i.e., intervention) to those who did not use the mDOT application (i.e., control). The investigators will compare medication adherence between intervention and control arms using the Medication Level Variability Index (MLVI), a validated measure of adherence derived from the standard deviation of measured drug levels (22-23).

   1.2 Secondary Objectives
   * Clinical endpoints including rejection and hospitalization
   * Patient reported adherence on immunosuppressant therapy instrument (ITAS)
   * Patient-reported QoL outcomes as measured by PedsQL and SF-36
   * Patient-reported self-efficacy using the Riekert Self-efficacy scale
   * Patient-reported usability using the PSSUQ (treatment arm only)
   * To examine the patterns of medication adherence in transplant recipients in both groups to better understand baseline medication adherence
   * To understand the feasibility and acceptability of implementing such a system into the clinical workflow and patient follow-up care management
2. BACKGROUND AND RATIONALE In adolescent and adult solid organ transplant recipients, poor adherence to immunosuppressant medications carries the risk of graft rejection, short- and long-term post-transplant complications, and increased healthcare costs (1-8). In transplant recipients, adherence to immunosuppressive drugs, as well as general medical indications is imperative to overall outcomes (9). The rate of non-adherence to immunosuppressive medications in transplant patients varies vastly, with reports ranging from 15-40% in adults and much higher at 50-70% among adolescents (9-14). Additionally, medication adherence is a key concern in the transition from adolescent to adult-centered transplant care, and transition planning should be prioritized in these transplant patients (15-18). Because of lacking objective and accurate non-adherence measurements, both to immunosuppressive drugs and medical indications, the true implications and prevalence of non-adherence is not yet well understood (19-21). Therefore, the investigators believe that mobile health (mHealth) technology has the potential to allow clinicians and researchers to more comprehensively address and understand non-adherence in adolescent and adult transplant recipients.

   emocha Mobile Health Inc. has developed an application that enables users to track dose-by-dose medication adherence through asynchronous, video directly observed therapy (DOT). This helps patients take medications as prescribed and gives providers the assurance that the patients are supported and successful in treatment. DOT is the practice of watching a patient take every dose of medicine in-person, and has typically only been done in extreme cases because it can be both costly and burdensome: DOT is the standard of care for Tuberculosis treatment and has proven high-adherence rates. Through mHealth technology, DOT can be used more broadly and without added burden; emocha's technology allows this through enabling patients to use the mobile application to view the regimen, record themselves taking every dose of the participant's medication, report side effects or symptoms, visualize treatment progress, and access educational content. This information is encrypted and transmitted to a HIPAA-secure web portal for providers to review. The aim of this study is to conduct a randomized control trial to compare medication adherence between patients who use the mHealth system against controls who do not.

   Emocha has formally evaluated the mDOT platform across several disease states: tuberculosis, Hepatitis C virus, and opioid use disorder. The U.S. Centers for Disease Control and Prevention (CDC) recognizes emocha's video modality as an acceptable form of DOT, according to the latest guidelines. To date, emocha has partnered with Johns Hopkins and three Maryland health department tuberculosis programs to assess quantitative, qualitative, and cost outcomes associated with emocha video DOT implementation. Among all participants - with more than 1,400 videos submitted thus far - mean patient adherence was 94 percent (median adherence 96 percent, interquartile range 93 to 100 percent). Similar adherence rates were proven in independent studies using emocha performed by Harris County, TX and the Puerto Rico Department of Health. Additionally, emocha is conducting a trial on the feasibility of video DOT for patients undergoing the initiation phase of buprenorphine treatment through office-based opioid treatment programs, as well as conducting ongoing research on Hepatitis C medication adherence among injection drug users.
3. STUDY DESIGN The purpose of this study is to understand how the use of an mHealth application, mDOT, changes medication adherence behaviors among liver or kidney transplant recipients. For the purpose of this research, the mobile app is a device of non-significant risk and exempt from the IDE requirement. emocha Mobile Health is the device manufacturer.

In this multi-center study, patients >/= 13 years of age who receive a liver or kidney transplant at Johns Hopkins Hospital, University of Virginia Medical Center or University of Miami Medical Center will be recruited to participate in this randomized control trial (RCT). There will be 2 arms participants may be randomly assigned to: intervention and control arms. Participants in the intervention arm will receive the mDOT application, and participants in the control arm will not. Both arms will still receive standard of care post-transplant.

Participants are followed for compliance with standard of care recommendations. No additional care or procedures will be administered to study participants. Given the uncertainty in whether this mHealth intervention will improve rates of immunosuppression medication adherence in liver and kidney transplant recipients, a non-treatment group is necessary in order to identify whether an advantage exists.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to participate in this study:

> 13 years old Own a smart phone and are willing to receive information through it Received a liver or kidney transplant at a participating study site during or prior to the study period.

Exclusion Criteria:

All candidates meeting any of the following exclusion criteria at baseline will be excluded from study participation:

Patients with cognitive impairments will not be eligible for enrollment due to inability to provide informed consent.

Inability or unwillingness of individual or legal guardian/representative to give consent.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cozumel Pruette, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 75 enrolled patients, however 5 dropped out before randomization and therefore only 70 were randomized to the arms.
Period: Overall Study
Arm/Group | mHealth Intervention | Standard of Care
Started | 36 | 34
Completed | 36 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Seventy participants recruited from 2 academic sites were enrolled in a pilot randomized controlled trial of mDOT for transplantation compared to standard-of-care in SOT participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | mHealth Intervention | Standard of Care | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 30 | 28 | 58
  >=65 years | 3 | 3 | 6
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.5 [21 to 75] | 44 [21 to 75] | 48.5 [23 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 34
  Male | 15 | 21 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 35 | 32 | 67
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 9 | 18
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 34 | 70
Nonadherence to immunosuppressant medication [Count of Participants; unit: Participants] — Baseline measure of adherence obtained from EMR documentation
  Participants
    Non-adherent | 0 | 1 | 1
    Adherent | 36 | 33 | 69

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence Via Medication Level Variability Index (MLVI)
Description: To compare medication adherence of solid organ transplant recipients, specifically liver and kidney transplants, using the mobile DOT (mDOT) application (i.e., intervention) to those who did not use the mDOT application (i.e., control). The investigators will compare medication adherence between intervention and control arms using the Medication Level Variability Index (MLVI), a validated measure of adherence derived from the standard deviation of measured drug levels. The investigators will look at the difference in MLVIs between the two solid organ transplant groups. MLVI is the standard deviation of a series of at least three trough blood levels of tacrolimus or sirolimus. Higher MLVI value indicates greater variability in medication levels. MLVI >=2 is suggestive of nonadherence and MLVI <2 suggestive of adherence.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | mHealth Intervention | Standard of Care
Number analyzed (Participants) | 36 | 34
Participants
  MLVI >=2 | 23 | 24
  MLVI <2 | 10 | 8
  Missing | 3 | 2

2. Secondary Outcome: Blood Tacrolimus Levels
Description: Clinical endpoint measuring the blood levels of tacrolimus (in ng/ml) that indicate rejection of transplant or not
Time Frame: 3 months
Measure: Median (Standard Deviation); unit: ng/ml
Arm/Group | mHealth Intervention | Standard of Care
Number analyzed (Participants) | 36 | 34
ng/ml | 2.6 (0.87) | 2.37 (1.07)

3. Secondary Outcome: Patient Reported Adherence
Description: Patient reported adherence depending on their scores from the immunosuppressant therapy instrument (ITAS questionnaire) will be measured. The ITAS is a four-item questionnaire that asks respondents to indicate how often they were non-adherent to immunosuppressant therapy (IST) given a particular circumstance. They are asked how often they: (i) forgot to take their IST medications; (ii) were careless about taking their IST medications; (iii) stopped taking their IST medications because they felt worse; and (iv) missed taking their IST medications for any reason. This is a binary measure where A stands for 0% of the time (none), B stands for 1%-20% of the time, C stands for 21-50% of the time, D stands for greater than 50% of the time. ITAS scores range from 0 to 12; 0 is the lowest score and 12 is the highest score, indicating perfect adherence.
Time Frame: 3 months
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | mHealth Intervention | Standard of Care
Number analyzed (Participants) | 36 | 34
score on a scale | 12 (2) | 11 (2)

4. Secondary Outcome: Patient Reported QoL as Assessed by the PedsQL
Description: Patient-reported QoL outcomes as measured by PedsQL to measure quality of life and medication adherence. Items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life).
Time Frame: 12 months
Population: Data not collected
Arm/Group | mHealth Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: mHealth Usability Measurement
Description: Patient-reported usability measured using the Post-Study System Usability Questionnaire (PSSUQ), a 16-item questionnaire that follows a 7-point Likert Scale. The scale starts with 1 (strongly agree) and ends with 7 (strongly disagree). The overall result is calculated by averaging the scores from the 7 points of the scale, for all 16 items. The lower the score, the better the usability and satisfaction. Median likert scale choice is reported. This will be done in the mHealth intervention arm only.
Time Frame: 3 months
Population: Three month assessment of all participants who completed the survey.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | mHealth Intervention
Number analyzed (Participants) | 15
score on a scale | 1.57 (1.47)

6. Secondary Outcome: Patterns of Medication Adherence
Description: To examine the patterns of medication adherence in transplant recipients in both groups to better understand baseline medication adherence. We will be doing this by looking at the adherence streaks (number of doses taken over number of doses expected).
Time Frame: 12 months
Population: Data not collected
Arm/Group | mHealth Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Provider Workflow as Assessed by Patient Usage of the mDOT App
Description: Provider clinical workflow will be measured by evaluating patient usage on the app.
Time Frame: 12 months
Population: Data not collected
Arm/Group | mHealth Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Patient Reported QoL as Assessed by the SF-36
Description: Patient Reported QoL Short Form (SF)-36 to measure quality of life and medication adherence. The scoring is scaled at 0 as the lowest and 100 as the highest. The lower the score, the more disability.
Time Frame: 12 months
Population: Data not collected
Arm/Group | mHealth Intervention | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | mHealth Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34

LIMITATIONS AND CAVEATS:
Challenges with recruitment in the setting of COVID pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT04587024/Prot_SAP_000.pdf